CLINICAL TRIAL: NCT01727245
Title: The Role of Adipose Tissue in Atherogenic Conditions in Man - Mechanisms and Interventions
Brief Title: NEFA (Non Esterified Fatty Acid) , Adipose Factors Behind Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Danderyd Hospital (Other); Ersta Hospital, Sweden (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Erik Näslund, Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011/1002-31/1
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Non-obese Controls
MeSH Terms: conditions — Obesity | interventions — Adiposity; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese (Other): Obese patients undergoing gastric by-pass surgery
  Interventions: Other: Obese
- Control group (Other): Cholecystectomy and anti-reflux surgery
  Interventions: Other: Control group

INTERVENTIONS:
Other: Obese — gastric bypass
  Arms: Obese
Other: Control group — Cholecystectomy and anti-reflux surgery
  Arms: Control group

SUMMARY:
We want to asses the role of adipose tissue for metabolic complications to obesity before and after weight loss (surgery).

ELIGIBILITY:
Inclusion Criteria obese:

* Bariatric surgery with laparoscopic gastric by-pass

Exclusion Criteria obese:

* diabetes mellitus typ 2 with insulin treatment and/or glitazones
* oral or parenteral steroid treatment
* complicated psychiatric disease
* Warfarin use

Inclusion Criteria non-obese controls:

* BMI under 30

Exclusion Criteria non-obese controls:

* diabetes
* oral or parenteral steroids treatment
* complicated psychiatric disease
* Warfarins use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity, adipose tissue function and gene function | two years after surgery
  Performed with hyperinsulinemic euglycemic clamp before and two years after surgery. Subcutaneous and visceral fat biopsy at the time of surgery.

SECONDARY OUTCOMES:
Body composition | two years after surgery
  DEXA (Dual-Energy X-ray absorptiometry), before and two years after surgery
Vascular function | two years after surgery
  Non invasive ultrasound of vascular stiffness, before and two years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Erik Näslund, Prof., Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Ersta Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Danderyds Hospital, Stockholm

REFERENCES:
- [Derived] Mileti E, Kwok KHM, Andersson DP, Mathelier A, Raman A, Backdahl J, Jalkanen J, Massier L, Thorell A, Gao H, Arner P, Mejhert N, Daub CO, Ryden M. Human White Adipose Tissue Displays Selective Insulin Resistance in the Obese State. Diabetes. 2021 Jul;70(7):1486-1497. doi: 10.2337/db21-0001. Epub 2021 Apr 16. PMID 33863803
- [Derived] Backdahl J, Andersson DP, Eriksson-Hogling D, Caidahl K, Thorell A, Mileti E, Daub CO, Arner P, Ryden M. Long-Term Improvement in Aortic Pulse Wave Velocity After Weight Loss Can Be Predicted by White Adipose Tissue Factors. Am J Hypertens. 2018 Mar 10;31(4):450-457. doi: 10.1093/ajh/hpx201. PMID 29177471